CLINICAL TRIAL: NCT03789487
Title: Prospective Multicentric Study of Electrical Optimization of Cardiac Resynchronization Therapy in Non-responder Patients
Brief Title: Electrical Optimization of Cardiac Resynchronization Therapy in Non-responder Patients
Acronym: OPTIREG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the end of inclusion period
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/09
Record Dates: First submitted 2018-12-17; First posted 2018-12-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Cardiac Resynchronization Therapy; Non-responders; Pacing vector optimization; Atrioventricular delay optimization; Non invasive hemodynamic optimization; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-responders to CRT (Experimental): Non-responders to CRT who will undergo an electrical optimization of the settings of their device
  Interventions: Device: Device programming of CRT pacemaker or defibrillator

INTERVENTIONS:
Device: Device programming of CRT pacemaker or defibrillator — Stimulation vector optimization then AV delay optimization in order to obtain the highest systolic blood pressure (SBP) by using the Finapress® NOVA noninvasive device

SUMMARY:
Cardiac Resynchronization Therapy (CRT) is an established treatment for patients with systolic heart failure and bundle branch block, improving functional capacity, quality of life and reducing morbi-mortality. However, one-third of patients are non-responders. Among factors associated with non-response, suboptimal electrical settings of the device, i.e. inadequate pacing vector selection and atrioventricular (AV) delay, is an important cause.

The aim of the study is to investigate whether the optimization of CRT settings (pacing vector and AV delay) results in improved clinical and echocardiographic outcomes in a non-responder CRT population after 6 months of therapy.

DETAILED DESCRIPTION:
This study is non-randomized, prospective, interventional, multicentric study. Patients who have been implanted with a CRT device between 6 and 18 months prior to inclusion and are considered non-responders are eligible for this study. CRT non-response can be clinical (lack of functional improvement or hospitalization for heart failure) and/or echocardiographic (insufficient improvement of LVEF and/or reduction of LVESV). Among exclusion criteria, permanent atrial fibrillation is of note.

Recruited patients will be submitted to an optimization procedure of their CRT device settings. This will be performed with a non-invasive method using the Finapress NOVA device, which records blood pressure with a digital cuff. The peak of blood pressure will correspond to the optimal device settings. The first step will be to chose the best pacing vector. The second step will be to chose the best AV delay. The best setting, i.e. associated with the highest blood pressure, will be programmed at the end of the optimization protocol.

The patients will be followed at 6 months with clinical evaluation and echocardiography to assess the conversion rate of non-responders to responders.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18
* Patient implanted with a CRT (CRT-P or CRT-D) more than 6 months but less than 18 months before inclusion
* Non-responder patients:

Clinical criteria (Packer classification):

Lack of improvement of NYHA functional class And/or hospitalization for heart failure

Echocardiographic criteria:

Lack of improvement of LVEF > 5points And/or reduction of LVESV < 15%

* Patient who had signed an informed consent and is willing to comply with study requirements
* Patient covered by French national healthcare insurance

Exclusion Criteria:

* Permanent/persistant atrial fibrillation/ supra-ventricular tachycardia
* Scheduled hospitalization for major cardiac intervention or cardiac surgery in the 6 coming months
* Life-expectancy of less than 6 months
* Pregnant or breastfeeding women
* Adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response | During the optimization session
  Highest Systolic Blood Pressure (SBP) obtained by stimulation vector

SECONDARY OUTCOMES:
echocardiographic response | at 6 months of follow-up
  Left Ventricular Ejection Fraction (LVEF), Left Ventricular end-diastolic Volume (LVEDV), Left Ventricular End-Systolic Volume (LVESV)
Clinical response | at 6 months of follow up
  Hospitalization for heart failure

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - GHEM Eaubonne, Montmorency
  - CHU de Poitiers, Poitiers
  - CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No